CLINICAL TRIAL: NCT04451291
Title: DSC-COVID-19: An Open-label Study on the Safety and Efficacy of Decidual Stromal Cells in Respiratory Failure Induced by COVID-19
Brief Title: Study of Decidual Stromal Cells to Treat COVID-19 Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-DEPLOY: DSC-COVID-19; 20-5527 (Other: University Health Network)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decidual Stromal Cells (DSC) (Experimental): Participants will receive one dose of DSC at 1x10^6/kg. A second dose may be given sometime between Day 5 and Day 8 if the participant's condition improves.
  Interventions: Biological: Decidual Stromal Cells (DSC)

INTERVENTIONS:
Biological: Decidual Stromal Cells (DSC) — DSCs are involved in the immune system during pregnancy. The DSCs used in this study will come from laboratory grown allogeneic human decidual stromal cells obtained from donated placentas.

SUMMARY:
This is a research study to see how safe and effective decidual stromal cells are in treating patients with respiratory failure (breathing problem where not enough oxygen is passed from the lungs into the blood) caused by COVID-19.

DETAILED DESCRIPTION:
COVID-19 viral infectious disease that has lead to high numbers of critically ill patients or death due to respiratory failure.

Decidual Stromal Cells (DSC) may be useful in the treatment of acute respiratory distress syndrome (ARDS) by reducing lung inflammation and then time that patients require help with breathing (mechanical ventilation).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent for participation in the study, either by the participant themselves or by the legally acceptable representative (LAR)
* Virological diagnosis of SARS-CoV-2 infection (PCR)
* Acute respiratory distress syndrome (ARDS) not due to cardiac causes
* Receiving mechanical ventilation

Exclusion Criteria:

* Severe comorbidity with life expectancy <3 months according to investigators assessment
* Currently receiving extracorporeal membrane oxygenation (ECMO)
* Patients with established positive bacterial blood cultures prior to enrollment or suspicion of superimposed bacterial pneumonia
* Patients with diagnosed significant pulmonary embolism or deep vein thrombosis in the previous 3 months
* Patients who have been intubated for more than 48 hours
* Known hypersensitivity to dimethyl sulfoxide (DMSO) or to porcine or bovine proteins
* Acute co-morbidity within 7 days before inclusion such as stroke
* History of severe chronic history of heart disease, recent myocardial infarction or unstable angina, lung disease (requiring home oxygen), pulmonary hypertension, or liver comorbidities
* Malignancy that requires treatment in the previous two years (excluding non-melanoma skin malignancies treated by excision, or cryotherapy)
* History of immunosuppression (immunomodulators or anti-rejection drugs in past year, or active disease, autoimmune disease on treatment, transplant recipients) or anaphylaxis
* Refusal of blood products
* Severe co-morbidity/co-morbidities which in the opinion of the investigators would compromise safety assessments
* Pregnant or breast-feeding
* Actively participating on another trial of an investigational agent for ARDS
* Unacceptable laboratory blood tests for alanine aminotransferase (ALT)/aspartate aminotransferase (AST), neutrophils, or platelets

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Number of ventilator free days following infusion of decidual stromal cells | 28 days

SECONDARY OUTCOMES:
Mortality rate from COVID-19 | 28 days
Mortality rate from COVID-19 | 60 days
Mortality rate from COVID-19 | 180 days
All-cause morality rate | 28 days
All-cause morality rate | 60 days
All-cause morality rate | 180 days
Average number of days in ICU | 180 days
Average number of days of hospital admittance | 180 days
Average days not requiring vasopressors | 180 days
Overall survival rate | 180 days
Average viral clearance | 180 days
Average number of days of supplemental oxygenation | 180 days
Average number of day without supplemental oxygen | 180 days
Mean PaO2/FiO2 as compared to patient baseline | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: John Granton, M.D., Principal Investigator — Toronto General Hospital
Locations (3):
- Canada (3):
  - Brampton Civic Hospital, Brampton, Ontario
  - Etobicoke General Hospital, Etobicoke, Ontario
  - Toronto General Hospital, Toronto, Ontario